CLINICAL TRIAL: NCT05091229
Title: A Cohort Study to Evaluate a Blood Test for Early-screening of Kawasaki Disease
Brief Title: A Blood Test to Diagnose Kawasaki Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: HBI Solutions Inc. (Industry)
Collaborators: Shanghai Children's Medical Center (Other); mProbe Inc. (Industry)
Responsible Party: Principal Investigator, Hao Zhang, Professor, HBI Solutions Inc.
Other Study IDs: KD_001
Record Dates: First submitted 2021-10-12; First posted 2021-10-25 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Kawasaki Disease
MeSH Terms: conditions — Mucocutaneous Lymph Node Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort A: Blood specimen collection. Study samples must be collected prior to any treatment.
- Cohort B: Blood specimen collection. Study samples must be collected prior to any treatment.
- Cohort C: Blood specimen collection. Study samples must be collected prior to any treatment.

SUMMARY:
A case-control cohort study is being conducted to develop and validate the performance of a whole blood gene expression qPCR test to distinguish KD from other febrile conditions by collecting whole blood sample from KD patients in the first 7 days of illness and from febrile controls immediately after presentation and before clinical diagnosis is confirmed.

DETAILED DESCRIPTION:
Currently, there is no diagnostic tool for Kawasaki disease (KD). Diagnosis is based on clinical features shared with other febrile conditions, frequently resulting in delayed or missed treatment and an increased risk of coronary artery aneurysms. An accurate diagnostic blood test might enable early discrimination of Kawasaki disease from other infectious and inflammatory conditions, resulting in a precise clinical treatment to improves survival and quality of children's life. The purpose of this study is to develop and validate a blood-based assay for accurate diagnosis of KD in in the first 7 days of illness.

The study will collect blood samples from healthy patients with no recent history of fever or immunization and from febrile patients diagnosed with KD or other infectious and inflammatory diseases.

Three types of patients in this study:

Cohort A:

Children ages 6-60 months old who have been diagnosed with (or strong clinical suspicion for) KD by clinician. Blood samples must be collected before any treatment has been initiated.

Cohort B:

Children ages 6-60 months old with febrile conditions who have been diagnosed with other infections or inflammation by clinician. Blood samples must be collected before any treatment.

Cohort C:

Children ages 6-60 months old with no recent history of fever or immunization.

ELIGIBILITY:
COHORT A

Inclusion Criteria:

* 6- 60 months of age
* Diagnosed with possible Kawasaki disease (even if they do not fulfil the criteria below for Kawasaki disease) by the treating clinician based on the 2004 AHA guidelines
* Appropriate guardian of patients are able and willing to provide blood samples per protocol
* Appropriate guardian of patients are able to comprehend and willing to sign and date the written informed consent document(s) and any applicable medical record release documents for the study

Exclusion Criteria:

* Patient with comorbidities likely to influence gene expression, such as immunosuppressive treatments,
* Have a medical condition which, in the opinion of the investigator, should preclude enrollment into the study.
* Have participated or be currently participating in a clinical research study in which an experimental medication has been administered

COHORT B

Inclusion Criteria:

* 6- 60 months of age
* Diagnosed with febrile illness but without Kawasaki disease presentation criteria
* Appropriate guardian of patients are able and willing to provide blood samples per protocol
* Appropriate guardian of patients are able to comprehend and willing to sign and date the written informed consent document(s) and any applicable medical record release documents for the study

Exclusion Criteria:

* Patient with comorbidities likely to influence gene expression, such as immunosuppressive treatments,
* Have a medical condition which, in the opinion of the investigator, should preclude enrollment into the study.
* Have participated or be currently participating in a clinical research study in which an experimental medication has been administered

COHORT C

Inclusion Criteria:

* 6- 60 months of age
* no recent history of fever or immunization
* Appropriate guardian of patients are able and willing to provide blood samples per protocol
* Appropriate guardian of patients are able to comprehend and willing to sign and date the written informed consent document(s) and any applicable medical record release documents for the study

Exclusion Criteria:

* Patient with comorbidities likely to influence gene expression, such as immunosuppressive treatments,
* Have a medical condition which, in the opinion of the investigator, should preclude enrollment into the study.
* Have participated or be currently participating in a clinical research study in which an experimental medication has been administered

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of Kawasaki Disease | 4 weeks
  Diagnosis of KD in patients made by KD experts (pediatric infectious disease or pediatric rheumatologists) based on the 2004 AHA guidelines.

SECONDARY OUTCOMES:
Coronary artery status | 6 weeks
  Coronary artery status and Z-score (SD from the mean adjusted for body surface area) for patients with KD, will be recorded. Coronary artery status will be classified as normal (right coronary artery (RCA) and left anterior descending (LAD) Z-score always <2.5) or abnormal (RCA and/or LAD Z-score ≥2.5 within the first 6 weeks after diagnosis).
Coronary artery aneurysm | 6 weeks
  Echo findings with coronary artery aneurysm

CONTACTS AND LOCATIONS:
Overall Officials: Hao Zhang, M.D, Principal Investigator — Shanghai Children's Medical Center

IPD SHARING:
Plan to Share IPD: Undecided